CLINICAL TRIAL: NCT00862784
Title: An Open Label, Multicenter, Phase 2 Study Evaluating the Safety and Efficacy of IMC-1121B in Combination With 5-FU/FA and Oxaliplatin (Modified FOLFOX-6) as First-line Therapy in Patients With Metastatic Colorectal Cancer
Brief Title: A Study of IMC-1121B (Ramucirumab) in Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13897; 2008-004936-19 (EudraCT Number); CP12-0709 (Other: ImClone Systems); I4T-IE-JVBH (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-05

CONDITIONS: Colorectal Carcinoma
Keywords: Colorectal carcinoma; CRC; Colon Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Ramucirumab; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMC-1121B (ramucirumab) + mFOLFOX-6 (Experimental): This regimen will be repeated every 2 weeks until disease progression, unacceptable toxicity, or withdrawal.
  Interventions: Biological: IMC-1121B (ramucirumab); Drug: Oxaliplatin; Drug: Folinic acid; Drug: 5-FU

INTERVENTIONS:
Biological: IMC-1121B (ramucirumab) — 8 milligrams/kilogram (mg/kg) IMC-1121B (ramucirumab) infusions every 2 weeks
  Other Names: ramucirumab; LY3009806
Drug: Oxaliplatin — 85 milligrams/square meter (mg/m²) intravenous infusion over 2 hours on Day 1
Drug: Folinic acid — 400 mg/m² intravenous infusion over 2 hours on Day 1
Drug: 5-FU — 400 mg/m² intravenous bolus injection over 2-4 minutes, immediately following folinic acid infusion
Drug: 5-FU — 2400 mg/m² intravenous continuous infusion over 46 hours immediately following bolus 5-FU on Days 1 and 2

SUMMARY:
The purpose of this study is to test how long participants with colorectal cancer live without progressive disease when being treated with IMC-1121B (ramucirumab) and the modified FOLFOX-6 chemotherapy.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the progression-free survival (PFS) in participants with metastatic colorectal cancer when treated with the monoclonal antibody IMC-1121B (ramucirumab) in combination with the modified FOLFOX-6 [folinic acid (FA) + fluorouracil (5-FU) + oxaliplatin, mFOLFOX-6] chemotherapy regimen as first-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* The participant must have histologically confirmed adenocarcinoma of the colon or rectum that is locally-advanced or metastatic and unresectable
* The participant has at least one unidimensionally-measurable target lesion [≥ 2 centimeters (cm) with conventional techniques or ≥ 1 cm with spiral computed tomography (CT) scan or magnetic resonance imaging (MRI), as defined by Response Evaluation Criteria in Solid Tumors (RECIST)]; target lesion(s) must not lie within an irradiated area. Participants with locally advanced rectal carcinoma who have undergone previous radiation must have documented evidence of disease progression in the pelvis in order to participate
* The participant is age ≥ 18 years
* The participant has a life expectancy of ≥ 6 months
* The participant has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-1 at study entry
* The participant has adequate hematologic function, as evidenced by an absolute neutrophil count (ANC) ≥ 1500/microliter (μL), hemoglobin ≥ 10 grams/deciliter (g/dL), and platelets ≥ 100,000/μL
* The participant has adequate hepatic function as defined by: total bilirubin ≤ 1.5 x upper limit of normal (ULN), aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 x ULN (or 5.0 x ULN in the case of liver metastases), and serum albumin ≥ lower limit of normal (LLN) institutional range or (if < LLN) within 10% of the LLN
* The participant has adequate renal function as defined by a serum creatinine ≤ 1.5 x ULN, or creatinine clearance (measured via 24-hour urine collection) ≥ 60 milliliters/minute (mL/min)
* The participant's urinary protein ≤ 1+ on dipstick or routine urinalysis [(UA); if urine dipstick or routine analysis is ≥ 2+, a 24-hour urine for protein must demonstrate < 1000 milligrams (mg) of protein in 24 hours to allow participation in the study]
* The participant must have adequate coagulation function as defined by International Normalized Ratio (INR) ≤ 1.5 and a partial thromboplastin time (PTT) ≤ 5 seconds above the ULN. Participants on full-dose anticoagulation must be on a stable dose of oral anticoagulant or low molecular weight (LMW) heparin and if on warfarin, must have an INR between 2 and 3 and no active bleeding or pathological condition present that carries a high risk of bleeding (for example, tumor involving major vessels or known varices)
* The participant has resolution to Grade ≤ 1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 3 (NCI-CTCAE v 3.0) of all clinically significant toxic effects of prior chemotherapy, surgery, radiotherapy, or hormonal therapy with the exception of peripheral neuropathy which must have resolved to Grade 0
* The participant agrees to use adequate contraception during the study period and for 8 weeks after the last dose of study treatment
* The participant has provided signed informed consent

Exclusion Criteria:

* The participant has received prior systemic chemotherapy for locally-advanced unresectable or metastatic colorectal cancer (CRC). Prior adjuvant chemotherapy is allowed if disease progression has been documented > 6 months after the end of the last cycle of adjuvant chemotherapy or > 12 months after the end of the last cycle of adjuvant oxaliplatin-containing regimens
* The participant has documented and/or symptomatic brain or leptomeningeal metastases
* The participant has participated in clinical studies of non-approved experimental agents or procedures within 12 weeks of study entry
* The participant has received previous therapy with monoclonal antibodies
* The participant has received previous therapy with any agent that targets vascular endothelial growth factor (VEGF) or VEGF receptor-2 (VEGFR-2) (including multi-targeted tyrosine kinase inhibitors)
* The participant has an ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia, psychiatric illness/social situations, or any other serious uncontrolled medical disorders in the opinion of the investigator
* The participant is on chronic non-topical corticosteroid treatment for > 6 months at doses > 10 mg/day of prednisolone or equivalent before study entry, which in the opinion of the investigator could compromise the participant or the study
* The participant has a known dihydropyrimidine dehydrogenase (DPD) deficiency
* The participant has a known allergy to any of the treatment components
* The participant has an acute or subacute intestinal obstruction
* The participant has uncontrolled or poorly controlled hypertension on a standard regimen of anti-hypertensive therapy
* The participant has a concurrent active malignancy other than adequately treated nonmelanomatous skin cancer, other noninvasive carcinoma, or in situ neoplasm. A participant with previous history of malignancy is eligible, provided that he/she has been disease free for > 3 years
* The participant, if female, is pregnant
* Has had prior autologous or allogeneic organ or tissue transplantation
* Has interstitial pneumonia or interstitial fibrosis of the lung, which in the opinion of the investigator could compromise the participant or the study
* Has pleural effusion or ascites that causes > Grade 1 dyspnea
* Has psychological, familial, sociological, or geographical conditions which do not permit adequate study follow-up, compliance with the protocol, or signature of Informed Consent
* Has undergone major surgery within 28 days prior to the first dose of study medication, or subcutaneous venous access device placement within 7 days prior to the first dose of study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- Canada (3):
  - ImClone Investigational Site, Ottawa, Ontario
  - ImClone Investigational Site, Toronto, Ontario
  - ImClone Investigational Site, Montreal, Quebec
- Spain (4):
  - ImClone Investigational Site, Barcelona
  - ImClone Investigational Site, Santander
  - ImClone Investigational Site, Seville
  - ImClone Investigational Site, Valencia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completer was defined as any participant who died due to any cause or progression of disease, or any participant who was alive and on study but off study treatment at the conclusion of the study.
Groups:
- IMC-1121B (Ramucirumab) + mFOLFOX-6: Received IMC-1121B (ramucirumab) 8 milligrams/kilogram (mg/kg) on Day 1 administered intravenously over 60 minutes and followed by administration of the modified FOLFOX-6 [folinic acid (FA) + fluorouracil (5-FU) + oxaliplatin, mFOLFOX-6] regimen as follows:
  Oxaliplatin 85 milligrams/square meter (mg/m²) intravenous infusion over 2 hours on Day 1; FA 400 mg/m² intravenous infusion over 2 hours on Day 1; 5-FU 400 mg/m² intravenous bolus injection over 2 to 4 minutes, immediately following the FA infusion; 5-FU 2400 mg/m² intravenous continuous infusion over 46 hours immediately following bolus 5-FU injection on Days 1 and 2.
  This regimen was repeated every 2 weeks until disease progression, unacceptable toxicity, or withdrawal.
Period: Overall Study
Arm/Group | IMC-1121B (Ramucirumab) + mFOLFOX-6
Started | 48
Received Any Amount of Study Drug | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who received any amount of study drug.
Arm/Group | IMC-1121B (Ramucirumab) + mFOLFOX-6
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 48
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 5
  Spain | 43

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from date of first dose to the first observation of progression of disease (PD) or death due to any cause. PD was determined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.0. PD is ≥20% increase in sum of longest diameter of target lesions and/or unequivocal progression of non-target lesion and/or new lesion. For participants who had no PD or death or had started new therapeutic anticancer treatment, PFS was censored at their last radiographic tumor assessment.
Time Frame: First dose to measured progressive disease or death due to any cause up to 28.1 months
Population: All participants who received any amount of study drug. The number of participants censored was 11.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMC-1121B (Ramucirumab) + mFOLFOX-6
Number analyzed (Participants) | 48
months | 11.5 [8.6 to 13.1]

2. Secondary Outcome: Percentage of Participants With Complete Response or Partial Response [Objective Response Rate (ORR)]
Description: ORR is the percentage of participants with a confirmed complete response (CR) + partial response (PR), as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.0. CR is disappearance of all target and non-target lesions; PR is a ≥30% decrease in sum of longest diameter of target lesions without new lesion and progression of non-target lesion. ORR is calculated as a total number of participants with CR or PR from the start of study treatment until disease progression or recurrence divided by the total number of participants treated, then multiplied by 100.
Time Frame: First dose to date of objective progressive disease up to 23.8 months
Population: All participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMC-1121B (Ramucirumab) + mFOLFOX-6
Number analyzed (Participants) | 48
percentage of participants | 58.3 [43.21 to 72.39]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first dose to the date of death due to any cause. For participants who were alive or were lost to follow-up, OS was censored on the last date the participant was known to be alive.
Time Frame: First dose to death due to any cause up to 28.1 months
Population: All participants who received any amount of study drug. The number of participants censored was 18.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMC-1121B (Ramucirumab) + mFOLFOX-6
Number analyzed (Participants) | 48
months | 20.4 [18.5 to 25.1]

4. Secondary Outcome: Duration of Response
Description: The duration of response was defined as the time from first objective status assessment of complete response (CR) or partial response (PR) to the first time of progression or death as a result of any cause. CR or PR is classified by the investigators according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.0. CR is disappearance of all target and non-target lesions; PR is a ≥30% decrease in sum of longest diameter of target lesions without new lesion and progression of non-target lesion.
Time Frame: Time of response to time of measured progressive disease up to 22.2 months
Population: All participants who received any amount of study drug who had CR and PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMC-1121B (Ramucirumab) + mFOLFOX-6
Number analyzed (Participants) | 28
months | 11.0 [6.9 to 12.6]

5. Secondary Outcome: Number of Participants With IMC-1121B (Ramucirumab)-Related Adverse Events (AEs)
Description: Data presented are the number of participants who experienced AEs of any grade and AEs of Grade ≥3 based on National Cancer Institute Common Terminology Criteria for Adverse Events, Version 3.0 (NCI-CTCAE v 3.0), that were considered to be related to IMC-1121B (ramucirumab) by the investigators. A summary of serious AEs (SAEs) and all other non-serious AEs regardless of causality, is located in the Reported Adverse Events module.
Time Frame: First dose to 25.2 months
Population: All participants who received at any amount of study drug.
Measure: Number; unit: participants
Arm/Group | IMC-1121B (Ramucirumab) + mFOLFOX-6
Number analyzed (Participants) | 48
participants
  Related AEs | 45
  Related AEs of Grade ≥3 | 19
  Related AE resulting in death | 2
  Related AE leading to discontinuation | 11

6. Secondary Outcome: Number of Participants With IMC-1121B (Ramucirumab)-Related Severe Adverse Events (SAEs)
Description: Data presented are the number of participants who experienced SAEs, adverse events (AEs) resulting in death and AEs leading to discontinuation of treatment, that were considered to be related to IMC-1121B (ramucirumab) by the investigators. A summary of SAEs and all other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: First dose to 25.2 months
Population: All participants who received any amount of study drug.
Measure: Number; unit: participants
Arm/Group | IMC-1121B (Ramucirumab) + mFOLFOX-6
Number analyzed (Participants) | 48
participants | 10

7. Secondary Outcome: Maximum Concentration (Cmax) at Day 1 of Cycle 1
Description: Due to sparse pharmacokinetic schedule, Cmax was not calculated.
Time Frame: Baseline, 1, 168, and 336 hours post infusion on Day 1 (Cycle 1)
Population: No participants were analyzed due to sparse pharmacokinetic schedule.
Arm/Group | IMC-1121B (Ramucirumab) + mFOLFOX-6
Number analyzed (Participants) | 0

8. Secondary Outcome: Area Under the Concentration (AUC) at Day 1 of Cycle 1
Description: Due to sparse pharmacokinetic schedule, AUC was not calculated.
Time Frame: Baseline, 1, 168, and 336 hours post infusion on Day 1 (Cycle 1)
Population: No participants were analyzed due to sparse pharmacokinetic schedule.
Arm/Group | IMC-1121B (Ramucirumab) + mFOLFOX-6
Number analyzed (Participants) | 0

9. Secondary Outcome: Half-Life (t1/2) at Day 1 of Cycle 1
Description: Due to sparse pharmacokinetic schedule, t1/2 was not calculated.
Time Frame: Baseline, 1, 168, and 336 hours post infusion on Day 1 (Cycle 1)
Population: No participants were analyzed due to sparse pharmacokinetic schedule.
Arm/Group | IMC-1121B (Ramucirumab) + mFOLFOX-6
Number analyzed (Participants) | 0

10. Secondary Outcome: Clearance (CL) at Day 1 of Cycle 1
Description: Due to sparse pharmacokinetic schedule, CL was not calculated.
Time Frame: Baseline, 1, 168, and 336 hours post infusion on Day 1 (Cycle 1)
Population: No participants were analyzed due to sparse pharmacokinetic schedule.
Arm/Group | IMC-1121B (Ramucirumab) + mFOLFOX-6
Number analyzed (Participants) | 0

11. Secondary Outcome: Steady State Volume of Distribution (Vss) at Day 1 of Cycle 1
Description: Due to sparse pharmacokinetic schedule, Vss was not calculated.
Time Frame: Baseline, 1, 168, and 336 hours post infusion Day 1 (Cycle 1)
Population: No participants were analyzed due to sparse pharmacokinetic schedule.
Arm/Group | IMC-1121B (Ramucirumab) + mFOLFOX-6
Number analyzed (Participants) | 0

12. Secondary Outcome: Maximum Concentration (Cmax) at Day 1 of Cycles 5, 9, 13, 17, and 21
Description: Due to sparse pharmacokinetic schedule, Cmax was not calculated.
Time Frame: Baseline and 1 hour post infusion on Day 1 (Cycles 5, 9, 13, 17, and 21)
Population: No participants were analyzed due to sparse pharmacokinetic schedule.
Arm/Group | IMC-1121B (Ramucirumab) + mFOLFOX-6
Number analyzed (Participants) | 0

13. Secondary Outcome: Area Under the Concentration (AUC) at Day 1 of Cycles 5, 9, 13, 17, and 21
Description: Due to sparse pharmacokinetic schedule, AUC was not calculated.
Time Frame: Baseline and 1 hour post infusion on Day 1 (Cycles 5, 9, 13, 17, and 21)
Population: No participants were analyzed due to sparse pharmacokinetic schedule.
Arm/Group | IMC-1121B (Ramucirumab) + mFOLFOX-6
Number analyzed (Participants) | 0

14. Secondary Outcome: Half-Life (t1/2) at Day 1 of Cycles 5, 9, 13, 17, and 21
Description: Due to sparse pharmacokinetic schedule, t1/2 was not calculated.
Time Frame: Baseline and 1 hour post infusion on Day 1 (Cycles 5, 9, 13, 17, and 21)
Population: No participants were analyzed due to sparse pharmacokinetic schedule.
Arm/Group | IMC-1121B (Ramucirumab) + mFOLFOX-6
Number analyzed (Participants) | 0

15. Secondary Outcome: Clearance (CL) at Day 1 of Cycles 5, 9, 13, 17, and 21
Description: Due to sparse pharmacokinetic schedule, CL was not calculated.
Time Frame: Baseline and 1 hour post infusion on Day 1 (Cycles 5, 9, 13, 17, and 21)
Population: No participants were analyzed due to sparse pharmacokinetic schedule.
Arm/Group | IMC-1121B (Ramucirumab) + mFOLFOX-6
Number analyzed (Participants) | 0

16. Secondary Outcome: Steady State Volume of Distribution (Vss) at Day 1 of Cycles 5, 9, 13, 17, and 21
Description: Due to sparse pharmacokinetic schedule, Vss was not calculated.
Time Frame: Baseline and 1 hour post infusion on Day 1 (Cycles 5, 9, 13, 17, and 21)
Population: No participants were analyzed due to sparse pharmacokinetic schedule.
Arm/Group | IMC-1121B (Ramucirumab) + mFOLFOX-6
Number analyzed (Participants) | 0

17. Secondary Outcome: Serum Anti-IMC-1121B (Immunogenicity) at Day 1
Description: Data presented are the number of participants with treatment emergent anti-IMC-112B antibodies.
Time Frame: Day 1 (Cycles 1, 5, 9, and 30-day follow-up)
Population: All participants who received any amount of study drug and had serum Anti-IMC-1121B (ramucirumab) evaluated.
Measure: Number; unit: participants
Arm/Group | IMC-1121B (Ramucirumab) + mFOLFOX-6
Number analyzed (Participants) | 48
participants
  Cycle 1 (n=39) | 0
  Cycle 5 (n=33) | 2
  Cycle 9 (n=25) | 0
  30-day Follow-up (n=17) | 2

ADVERSE EVENTS:
Arm/Group | IMC-1121B (Ramucirumab) + mFOLFOX-6
Serious Adverse Events (participants affected / at risk) | 18/48
Other Adverse Events (participants affected / at risk) | 47/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | IMC-1121B (Ramucirumab) + mFOLFOX-6 (N=48)
COAGULOPATHY (Blood and lymphatic system disorders) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (3)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) — Event resulted in death and occurred within 30 days of last dose
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) — Event resulted in death and occurred within 30 days of last dose
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
DISEASE PROGRESSION (General disorders) | 2 (2)
PYREXIA (General disorders) | 2 (2)
ABDOMINAL ABSCESS (Infections and infestations) | 1 (1)
ANAL ABSCESS (Infections and infestations) | 1 (1)
HAEMOPHILUS INFECTION (Infections and infestations) | 1 (1)
PELVIC ABSCESS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
UROSEPSIS (Infections and infestations) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
NEPHROTIC SYNDROME (Renal and urinary disorders) | 1 (1)
OVARIAN TORSION (Reproductive system and breast disorders) | 1/23 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1)
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-1121B (Ramucirumab) + mFOLFOX-6 (N=48)
ANAEMIA (Blood and lymphatic system disorders) | 8 (12)
HAEMOGLOBINAEMIA (Blood and lymphatic system disorders) | 3 (3)
LEUKOPENIA (Blood and lymphatic system disorders) | 8 (22)
NEUTROPENIA (Blood and lymphatic system disorders) | 27 (101)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 17 (41)
CONJUNCTIVITIS (Eye disorders) | 4 (4)
ABDOMINAL PAIN (Gastrointestinal disorders) | 13 (14)
CONSTIPATION (Gastrointestinal disorders) | 10 (13)
DIARRHOEA (Gastrointestinal disorders) | 32 (150)
DYSPEPSIA (Gastrointestinal disorders) | 5 (7)
FLATULENCE (Gastrointestinal disorders) | 3 (3)
HAEMORRHOIDS (Gastrointestinal disorders) | 3 (3)
NAUSEA (Gastrointestinal disorders) | 21 (52)
PROCTALGIA (Gastrointestinal disorders) | 3 (6)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 4 (9)
STOMATITIS (Gastrointestinal disorders) | 8 (16)
VOMITING (Gastrointestinal disorders) | 12 (28)
ASTHENIA (General disorders) | 35 (154)
FATIGUE (General disorders) | 4 (10)
INFUSION RELATED REACTION (General disorders) | 9 (18)
MUCOSAL INFLAMMATION (General disorders) | 26 (61)
OEDEMA PERIPHERAL (General disorders) | 11 (19)
PYREXIA (General disorders) | 13 (22)
NASOPHARYNGITIS (Infections and infestations) | 5 (8)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (11)
URINARY TRACT INFECTION (Infections and infestations) | 5 (10)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 (6)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (6)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 5 (9)
WEIGHT DECREASED (Investigations) | 3 (3)
ANOREXIA (Metabolism and nutrition disorders) | 11 (15)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (6)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 (11)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (5)
DIZZINESS (Nervous system disorders) | 3 (3)
DYSAESTHESIA (Nervous system disorders) | 23 (97)
DYSGEUSIA (Nervous system disorders) | 7 (10)
HEADACHE (Nervous system disorders) | 7 (11)
HYPOAESTHESIA (Nervous system disorders) | 3 (10)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 5 (11)
NEUROTOXICITY (Nervous system disorders) | 32 (71)
PARAESTHESIA (Nervous system disorders) | 7 (12)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 5 (9)
INSOMNIA (Psychiatric disorders) | 4 (4)
DYSURIA (Renal and urinary disorders) | 3 (4)
HAEMATURIA (Renal and urinary disorders) | 3 (3)
PROTEINURIA (Renal and urinary disorders) | 6 (10)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (5)
DYSAESTHESIA PHARYNX (Respiratory, thoracic and mediastinal disorders) | 6 (8)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 4 (5)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 (7)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 15 (20)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 3 (4)
ALOPECIA (Skin and subcutaneous tissue disorders) | 9 (10)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 4 (5)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 4 (7)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 11 (22)
HYPERTENSION (Vascular disorders) | 27 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.